CLINICAL TRIAL: NCT04685343
Title: Behavioral and Neural Phenotypes of Primary Dysmenorrhea in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laura Payne, Assistant Professor, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P001729
Record Dates: First submitted 2020-12-02; First posted 2020-12-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fMRI and laboratory pain induction (Experimental)
  Interventions: Behavioral: Quantitative Sensory Testing; Other: fMRI

INTERVENTIONS:
Behavioral: Quantitative Sensory Testing — Quantitative sensory testing (QST) consisting of 4 pain induction and sensory sensitivity tasks (i.e., pressure applied to the thumbnail, arms, shoulders, and lower abdomen, a cold water task, and one video-watching task).
Other: fMRI — Functional magnetic resonance imaging (fMRI) session consisting of structural and functional brain scans.

SUMMARY:
The study will use primary dysmenorrhea (PD; menstrual pain without an identified organic cause) as a model to examine biomarkers associated with menstrual and non-menstrual bodily pain in adolescent girls, ages 13-19. Participants will undergo extensive phenotyping including pain inhibition testing and multimodal neuroimaging to obtain indices brain structure and function at baseline and 12 months later. Menstrual pain severity and non-menstrual bodily pain will be assessed monthly for 24 months. Aims of the study are: 1) to identify the central mechanisms of PD using measures of pain inhibition and brain structure and connectivity of sensorimotor, default, emotional arousal, and salience networks, 2) to determine deficits in pain inhibition and alterations in brain structure and network connectivity that predict the one-year developmental trajectories of menstrual pain and non-menstrual bodily pain, and 3) to identify the dynamic relationship between alterations in pain inhibition and brain structure and connectivity with symptom change in menstrual pain and non-menstrual bodily pain. We hypothesize that deficits in endogenous pain inhibition and alterations in brain structure, connectivity, and function of regional networks will be positively associated with menstrual pain severity ratings at baseline and predict the trajectory of menstrual and non-menstrual bodily pain over 2 years. The results are expected to identify specific mechanisms and characteristics that predict the transition from acute/cyclical pain to persistent or chronic pain, which will support the development of therapies to prevent the transition from recurrent to chronic pain in adulthood.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 13-19 years
2. Self-reported menstrual cycle averaging 22-35 days
3. Regular menstrual cycles for at least 6 months
4. Access to a smartphone or email
5. Right handed
6. Body Mass Index (BMI) of 35 or less
7. Able to read and understand English
8. Ability and willingness to provide written informed assent/consent
9. Availability of a parent to provide written parental permission (for participants under age 18)

Exclusion Criteria:

1. Use of oral contraceptives or any exogenous hormones in the previous 3 months prior to participation
2. Presence of factors indicative of secondary dysmenorrhea (e.g., self-reported presence of persistent pelvic pain throughout the month)
3. Diagnosis of chronic pain condition (e.g., Irritable bowel syndrome (IBS), functional abdominal pain, interstitial cystitis/painful bladder syndrome)
4. Current self-reported severe depression, bipolar disorder, panic disorder, or ADHD, or current treatment for these conditions
5. Diagnosis of an eating disorder within the last 6 months
6. Current or past diagnosis of any psychotic disorder
7. Currently pregnant
8. Self-reported weekly use of alcohol, cannabis, and/or other illegal substances
9. Use of stimulants (including methamphetamine and/or medications for the treatment of ADHD) or opioids in the previous 3 months. Participants who use other analgesics will be included but will be requested to not take these analgesics within the previous 24 hours of the laboratory session
10. History of pelvic inflammatory disease or sexually transmitted disease
11. Acute illness or injury that would potentially impact pain task performance (e.g., fever, flu symptoms) or that affect sensitivity of the extremities (e.g., Reynaud's disease). Potential participants who are being treated for cardiovascular disease(s) will be included pending discussion with the participant's primary physician
12. Developmental delay, diagnosis of autism, or significant cognitive impairment that may preclude understanding of study procedures
13. Presence of certain ferromagnetic appliance or implants (braces, retainers, spacers, wires, screws, etc.) in the mouth or any other body part that may be a contraindication for the magnetic resonance imaging (MRI) scanner
14. Significant fear of enclosed places (claustrophobia)

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Menstrual pain | Baseline
  Rating of average pain during the first two days of the most recent menstrual period on a 0 (no pain) to 10 (worst pain possible) numeric rating scale.
Change in menstrual pain from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Change in the rating of average pain during the first two days of the most recent menstrual period on a 0 (no pain) to 10 (worst pain possible) numeric rating scale.
Change in bodily pain from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Change in the number of bodily locations endorsed as painful during the prior month.
Pressure pain sensitivity (PPS) | At baseline
  The pain rating [on a 0 (no pain) to 100 (worst pain possible) numeric rating scale] of a 5-second, 2.0 kg/cm2 application of pressure to the right thumbnail bed.
Pressure pain tolerance (PPT) | At baseline
  The last rated pressure delivered in a series of increasing pressure applications to the right thumbnail bed. Each application of pressure lasts for 5 seconds. The pressure sequence is terminated when the participant reaches their individual tolerance and decides to stop, when the participant reaches the safety maximum amount of pressure, or when the participant rates the pressure >=80 on a 0 (no pain) to 100 (worst pain possible) numeric rating scale.
Trapezius pressure pain threshold (TPPTh) | At baseline
  The amount of pressure, applied by a pressure algometer to the participant's trapezius muscle, needed for the pressure stimulus to first feel painful to the participant.
Conditioned pain modulation (CPM) | At baseline
  Conditioned pain modulation (CPM) assesses pain inhibition. CPM is calculated as the change in the TPPTh between when the pressure is applied by itself (test stimulus) and when it is applied while the participant's hand is submerged in cold water (conditioning stimulus).
Gray matter volume | At baseline
  Gray matter regional volume and surface area will be measured from images obtained during the fMRI session.
White matter fiber tract values | At baseline
  Obtained from fiber tracking using images obtained during diffusion tensor imaging (DTI). Values represent anatomical connectivity of cortical and subcortical brain regions.
Resting state networks | At baseline
  Calculated from images obtained during resting state fMRI. Region-to-region connectivity indices are obtained by correlating fMRI time series corrected for physiological noise and motion. Region-to-region connectivity strength of the regions of interest (i.e., salience, sensorimotor, emotional arousal, and default mode networks) will be assessed for each participant.

SECONDARY OUTCOMES:
Change in menstrual pain from 12-months post baseline to 24-months post baseline | 12 months after baseline and 24 months after baseline
  Change in the rating of average pain during the first two days of the most recent menstrual period on a 0 (no pain) to 10 (worst pain possible) numeric rating scale.
Change in bodily pain from 12-months post baseline to 24-months post baseline | 12 months after baseline and 24 months after baseline
  Change in the number of bodily locations endorsed as painful during the prior month.
Salivary pro-inflammatory cytokines | Three time points during each of two study visits: during questionnaire completion (approx. 20 min. after arrival), immediately after the imaging session (approx. 90 min. after arrival), and following the final pain task (approx. 120 min after arrival)
  Assessment of pro-inflammatory cytokines found in the saliva (e.g., IL-1 Beta, IL-6, IL-8, TNF-Alpha)
Trapezius pressure pain threshold (TPPTh) | 12 months after baseline
  The amount of pressure, applied by a pressure algometer to the participant's trapezius muscle, needed for the pressure stimulus to first feel painful to the participant.
Change in conditioned pain modulation (CPM) from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Alterations in pain inhibition will be assessed via the direction of the change (i.e., improvement in pain inhibition, worsening of pain inhibition, and stable pain inhibition) as well as the magnitude of the change.
Change in pressure pain sensitivity (PPS) from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Change in the pain rating [on a 0 (no pain) to 100 (worst pain possible) numeric rating scale] of a 5-second, 2.0 kg/cm2 application of pressure to the right thumbnail bed.
Change in pressure pain tolerance (PPT) from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Change in the PPT described above between baseline and 12-months post baseline.
Change in gray matter volume from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Change in the gray matter regional volume and surface area obtained from images obtained during the fMRI session.
Change in white matter fiber tract values from baseline to 12-months post baseline | At baseline and 12 months after baseline
  Change in the DTI-produced fiber tracking values, which represent anatomical connectivity of cortical and subcortical brain regions.
Change in resting state networks | At baseline and 12 months after baseline
  Change in region-to-region connectivity strength of the regions of interest (i.e., salience, sensorimotor, emotional arousal, and default mode networks).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Payne, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Payne LA, Handy AB, Seidman LC, Mitchell CM, Edwards RR. Multisensory sensitivity predicts menstrual pain and widespread pain trajectories over 12 months in adolescents with and without primary dysmenorrhea. Pain. 2025 Nov 24. doi: 10.1097/j.pain.0000000000003868. Online ahead of print. PMID 41284472